CLINICAL TRIAL: NCT03166748
Title: Compare the Clinical/Radiographic Outcomes of Potassium Nitrate in Polycarboxylate Cement and MTA as Pulpotomy Biomaterials Used for Asymptomatic Vital Immature Permanent Lower First Molars
Brief Title: Clinical and Radiographic Assessments of Potassium Nitrate in Polycarboxylate Versus Mineral Trioxide Aggregate as Pulpotomy Biomaterials in Immature Mandibular First Permanent Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Ibrahim Ahmed, master candidate at endodontic department faculty of dentistry cu, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBC-CU-2017-0518
Record Dates: First submitted 2017-05-16; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Pulpotomy of Immature Lower First Molar(Apexegenesis)
Keywords: Incomplete lower first molar; Immature permanent molar; Potassium nitrate in polycarboxylate; Mineral trioxide aggregate .Mineral trioxid
MeSH Terms: interventions — potassium nitrate; Polycarboxylate Cement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTA pulpotomy (Active Comparator): mineral trioxide aggregates (MTA) is accepted as an optimum material for use in vital pulp therapy of permanent teeth
  Interventions: Combination Product: Potassium Nitrate in Polycarboxylate cement
- Potassium Nitrate in Polycarboxylate cement (Experimental): Potassium nitrate (KNO3) is a superior desensitizer for hypersensitive teeth. Used with polycarboxylate cement, it serves as an effective liner for deep carious lesions. Also when placed under deep restorations with less than 1 mm of protective dentin remaining, it was effective in preserving pulpal vitality and it diminished the incidence and severity of post-restoration pain. As temporary cement (Kno3/zinc oxide eugenol [ZOE]) It reduced pain following full crown preparation.
  Interventions: Combination Product: Potassium Nitrate in Polycarboxylate cement

INTERVENTIONS:
Combination Product: Potassium Nitrate in Polycarboxylate cement — The application of polycarboxylate cement containing 5% KNO3 for direct capping of traumatically exposed pulp in animal models did not result in any degenerative changes in dental pulp, thought creating optimal conditions for preservation of pulp vitality and root completion.
  Polycarboxylate cement has very thin film thickness and bonds firmly to the tooth structure, is capable of withstanding the overlying pressure during restoration procedures. The good adhesive properties of polycarboxylate cement containing 5% KNO3 guaranteed the closure of cavity, good and lasting protection of traumatically exposed dental pulp and the formation of alkaline environment possessing a strong antiacidic, anti-inflammatory and antibacterial effect of this pulp capping material, creating optimal conditions for expression of its natural reparative potential. The increased release of potassium nitrate from polycarboxylate cement by time, might be the cause of decreasing the inflammatory intensity

SUMMARY:
The purpose of this RCT is to compare the clinical/radiographic outcomes of Potassium nitrate in polycarboxylate cement and MTA as pulpotomy biomaterials used for asymptomatic vital immature permanent lower first molar and this will help to clinically evaluate the use of alternative capping material in vital pulpotomy in young permanent teeth with pathologic pulpal injuries emphasis is set on avoiding total pupectomy and maintaining radicular pulp vitality and function and therefore maintain the tooth in a viable condition that help root completion.

DETAILED DESCRIPTION:
introduction: Vital pulp therapy (VPT) is defined as a treatment which aims to preserve and maintain pulp tissue that has been compromised but not destroyed by caries, trauma, or restorative procedures in a healthy state. Pulpotomy is one of the techniques of VPT where unhealthy pulp in pulp chamber is amputated leaving the healthy one in radicular part in root canal. This is particularly important in the young adult tooth with incomplete apical root development.

An important benefit for preservation of vital pulp is the protective resistance to mastication forces compared with a root-canal-filled tooth. It is reported that the survival rate of endodontically treated teeth is not as good as vital teeth especially in molars.

VPT is primarily recommended to be performed in young patients because of the high healing capacity of pulp tissue compared to older patients. The presence of an adequate blood supply is required for the maintenance of the pulp vitality. In addition, the presence of a healthy periodontium is necessary for success of VPT, where teeth with moderate to severe periodontal disease are not suitable candidates for the treatment.The prognosis of VPT is significantly reduced in cases with inadequate coronal seal and subsequent bacterial microleakage.

One of the most important issues in VPT is the status of the pulp tissue. The traditional school of thought is that VPT should only be carried out in teeth with signs and symptoms of reversible pulpitis.

After amputation of coronal pulp tissues Control of hemorrhage is also necessary for the success of VPT. Various options are available for the achievement of pulp hemostasis such as mechanical pressure using a sterile cotton pellet which may be soaked in sterile water, sodium hypochlorite and saline. Cases with signs of prolonged bleeding for more than 5 minutes are not candidates for pulpotomy.

Ferric sulfate (Fe2 [SO4]3) solution, 15.5%, is used commonly as a hemostatic retraction agent for crown and bridge impressions. Ferric sulfate is proposed as a pulpotomy agent on the theory that its mechanism of controlling hemorrhage might minimize the chances for inflammation and internal resorption believed by some investigators (Schroeder). The mechanism of action of ferric sulfate is probably by agglutination of ferric ion proteins complex results from the reaction of blood with both the ferric and sulfate ions that occlude the capillary orifices.

An appropriate pulp-capping agent establishes a biologically acceptable environment for the pulp tissue and prevents future bacterial contamination. The material should be biocompatible, bactericidal, provide a biologic seal, and induce hard tissue formation.

For many decades, calcium hydroxide has been the material of choice amongst the various pulp capping materials that are available. Clinical studies have reported a high rate of favorable outcomes of partial pulpotomies carried out with calcium hydroxide in cariously exposed young permanent molars. Despite its common use, it has several disadvantages including the presence of tunnel defects in induced dentinal bridges, obliteration of root canals making future endodontic treatment difficult, poor adherence to dentine, soluble, degrades with time and lack of long-term seal.

Currently, mineral trioxide aggregates (MTA) is accepted as an optimum material for use in vital pulp therapy of permanent teeth. MTA successful clinical outcome is reported to be due mainly to its long-term sealing ability and the stimulation of a high quality and a great amount of reparative dentin. In human clinical trials carried out on cariously exposed permanent teeth, the success rate of vital pulp therapy using MTA was considered to be high and ranged from 93 to 100%.

Despite its many advantages, MTA has some drawbacks that include the presence of toxic elements in the material composition, difficult handling characteristics, long setting time , tooth discoloration , and high cost, thus is an alternative material to MTA as a pulpotomy agent would be highly recommended.

Potassium nitrate (KNO3) is a superior desensitizer for hypersensitive teeth. Used with polycarboxylate cement, it serves as an effective liner for deep carious lesions. Also when placed under deep restorations with less than 1 mm of protective dentin remaining, it was effective in preserving pulpal vitality and it diminished the incidence and severity of post-restoration pain (27). As temporary cement (Kno3/zinc oxide eugenol [ZOE]) It reduced pain following full crown preparation.

Interestingly, using Potassium Nitrate with Dimethyl Isosorbide and Polycarboxylate Cement proved to be an effective direct capping agent for carious exposed vital pulps.

Polycarboxylate cement has very thin film thickness and bonds firmly to the tooth structure, is capable of withstanding the overlying pressure during restoration procedures. The good adhesive properties of polycarboxylate cement containing 5% KNO3 guaranteed the closure of cavity, good and lasting protection of traumatically exposed dental pulp and the formation of alkaline environment possessing a strong antiacidic, anti-inflammatory and antibacterial effect of this pulp capping material, creating optimal conditions for expression of its natural reparative potential. The increased release of potassium nitrate from polycarboxylate cement by time, might be the cause of decreasing the inflammatory intensity due to its antimicrobial action.

The application of polycarboxylate cement containing 5% KNO3 for direct capping of traumatically exposed pulp in animal models did not result in any degenerative changes in dental pulp. In fact, polycarboxylate cement containing 5% KNO3 was recommended as a basis for clinical investigations as a direct capping material.

So the present study seeks to investigate the clinical usefulness of applying polycarboxylate cement containing 5% KNO3 as a pulpotomy agent material of exposed immature permanent molars, thought creating optimal conditions for preservation of pulp vitality and root completion.

Up to the author knowledge, no previous randomized clinical trials (RCT) have evaluated the use of polycarboxylate containing KNO3 as a pulpotomy material, presenting a knowledge gap regarding this point.

Methods:

Source of patients: Out patients of the clinic of pedodontic at the faculty of oral and dental medicine, Cairo University.

Medical and dental history, will be obtained from all patients participating in this research followed by a thorough clinical and radiographic examination of deep carious mandibular first molar with no signs of irrivirsable pulpitis.

Preoperative radiographs will be acquired by using the standardized paralleling technique with the Rinn XCP alignment system (Rinn Corporation, Elgin, IL). Periapical radiographs will digitized and measurement done via Image J software (ImageJ v1.44; National Institutes of Health, Bethesda, MD).

Grouping of participants

According to sample size calculation, figure 2, fifty patients will be equally divided according to randomization table in to two groups:

* Experimental group: patient will be treated with 5% potassium nitrate and carboxylate cement pulpotomy.
* Control group: patient will be treated with MTA pulpotomy. Procedure steps

  1. Anesthesia Patient will be anesthetized by using nerve block local anesthesia (Carpule Mepecaine-L, Alexandria Company for Pharmaceuticals and Chemical Industries, Egypt).
  2. Access cavity All caries will be removed and the pulp chamber will be accessed with sterile high speed carbide round bur and endo-z bur bur to reflect the internal anatomy of the pulp chamber, and to remove its roof, taking the exposure as a starting point. The teeth were isolated with a rubber dam. The pulps will be amputated with a sterile # 5 round bur or a sharp spoon excavator, producing minimal trauma. Bleeding will controlled by placing a sterile cotton pellet on the amputated pulp soaked in saline to achieve a complete hemostasis at this stage for success of pulpotomy agent.
  3. Control of bleeding Ferric sulfate 15.5% solution in a plastic syringe and a cotton-tipped needle (viscostat, ultradent products Inc, Salt Lake City, USA) as a hemostatic and preservative agent. A small amount of ferric sulfate will be applied by gently wiping the cotton tip of the needle against the amputated pulp for 15 sec., flushed from the pulp chamber with a saline in order to remove any pieces of blood clot formation, dried with sterile cotton pellet and the access cavity will be dressed with pulpotomy agent; either mineral trioxide aggregate (white MTA Angelus,londrina,pr,brazil) or 5% potassium nitrate in polycarboxylate cement.(potassiun nitrate (KNO3),Merck,Darmstadt,Germany) according to randomization.

In the control group (MTA), the cavity will be covered with white MTA. One gram of cement powder will be mixed with a premeasured unit dose of 0.3 mL distilled water to achieve a powder/liquid ratio of 3:1 as per manufacturer's instructions. After 30 seconds of mixing, a putty consistency was obtained with a working time of about 5 minutes. The mix will delivered to the pulp stumps with the help of an MTA applicator (Angelus, Londrina, Brazil) and condensed lightly with a moistened sterile cotton pellet to ensure a 3- to 4-mm thickness. Because the setting time of MTA is about 4 hours, the MTA mixture will covered with a moistened cotton pellet, and the cavity will temporized with Cavit (ESPE, Seefeld, Germany), radiographic image will be taken to assure the level of the material in canal orifices. The following day the patient will be recalled, the cotton pellet will be removed, and the coronal pulp chamber will be sealed with resin modified glass ionomer (prime dent, Chicago, USA). The cavity will be filled with composite as a permanent restoration.

In the intervention group (potassium nitrate in polycrboxylate) the cavity will covered with 5% potassium nitrate (powder) (potassiun nitrate (KNO3),Merck,darmstadt,germany) which will mixed with the polyacrylic acid (liquid) (SIMENT P,Deepak product, inc, florida, USA) in 1:1 P/L ratio according to manufacturer directions. The mixed material will placed in the access cavity and light pressure will applied with a wet cotton pellet to contact the material with the pulp tissue. And the cavity will temporized with Cavit (ESPE, Seefeld, Germany), radiographic image will be taken to assure the level of the material in canal orifices. The following day the patient will be recalled, the temporary filling will removed, and the coronal pulp chamber will sealed with resien modified glass ionomer(prime dent, chicago,usa) the cavity will sealed with resien modified glass ionomer(prime dent, chicago,usa). The cavity will then filled with composit as a permanent restoration.

The patient will recalled for clinical evaluations at five follow up periods, and radiographic evaluations four follow up periods.

In case of post operative emergency (pain and/or swelling) an emergency appointment will be scheduled and shift of treatment to total pulpectomy and total root canal treatment will be done.

* Outcome If the tooth will functional without signs ⁄symptoms of pulp and periradicular inflammation⁄ infection (including spontaneous pain, sensitivity to percussion ⁄ palpation, soft tissue swelling or sinus tract and excessive mobility) in each follow-up time (24hr post operative,1 week, 3 month, 6 and 12 months after treatment), the treatment will clinically considered a success.

If root maturegenesis is evident radiographically without signs of failure (including formation of periradicular ⁄ interradicular lesion, internal ⁄ external root resorption) in each follow- up time (3 month, 6 and 12 months after treatment), the treatment will radiographically considered a success.

Radiometric analysis will be done via measurements throw image J software to evaluate the change in root length, dentin thickness and apical diameter measurement via ImageJ software (ImageJ v1.44; National Institutes of Health, Bethesda, MD).

ELIGIBILITY:
Inclusion Criteria:

* Egyptian children from 6-9 years
* Pathological caries or traumatic exposure
* lower immature first molar
* Asymptomatic irreversible pulpitis (no clinical symptoms of tooth or periapical pain in case of deep dental caries with pulp exposure during caries excavation

Exclusion Criteria:

* -Case of necrotic pulp tissue
* Pulp polyp
* Tooth tender to percussion
* Clinical progression into abscess formation.
* Medically compromised patient
* Tooth with abnormal anatomy
* Furcation involvement or canal calcification
* Excessive bleeding from root canal
* Tooth is unrestorable

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
clinical signs and symptoms assessment | 1 week, 3 month, 6 and 12 months after treatment
  patient will take a chart to make yes or no in this cases spontaneous pain,
  sensitivity to percussion ⁄ palpation
  excessive mobility
  soft tissue swelling
  sinus tract

SECONDARY OUTCOMES:
radiographic assessment of root completion | post operative,3 month, 6 and 12 months after treatment)
  radiographic assessment of root completion using radiometric analysis will be used to evaluate change in root length and dentin wall thickness at the end of study by aids of image j soft ware

CONTACTS AND LOCATIONS:
Overall Officials: Ghada El Hilaly eid, Professor of Endodontics, Study Chair — operator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ward J. Vital pulp therapy in cariously exposed permanent teeth and its limitations. Aust Endod J. 2002 Apr;28(1):29-37. doi: 10.1111/j.1747-4477.2002.tb00364.x. PMID 12360679
- [Background] Cvek M. A clinical report on partial pulpotomy and capping with calcium hydroxide in permanent incisors with complicated crown fracture. J Endod. 1978 Aug;4(8):232-7. doi: 10.1016/S0099-2399(78)80153-8. No abstract available. PMID 283188
- [Background] Al-Hiyasat AS, Barrieshi-Nusair KM, Al-Omari MA. The radiographic outcomes of direct pulp-capping procedures performed by dental students: a retrospective study. J Am Dent Assoc. 2006 Dec;137(12):1699-705. doi: 10.14219/jada.archive.2006.0116. PMID 17138715
- [Background] Caplan DJ, Cai J, Yin G, White BA. Root canal filled versus non-root canal filled teeth: a retrospective comparison of survival times. J Public Health Dent. 2005 Spring;65(2):90-6. doi: 10.1111/j.1752-7325.2005.tb02792.x. PMID 15929546
- [Background] Ricketts D. Management of the deep carious lesion and the vital pulp dentine complex. Br Dent J. 2001 Dec 8;191(11):606-10. doi: 10.1038/sj.bdj.4801246. PMID 11770946
- [Background] Stanley HR. Pulp capping: conserving the dental pulp--can it be done? Is it worth it? Oral Surg Oral Med Oral Pathol. 1989 Nov;68(5):628-39. doi: 10.1016/0030-4220(89)90252-1. PMID 2682429
- [Background] Demarco FF, Rosa MS, Tarquinio SB, Piva E. Influence of the restoration quality on the success of pulpotomy treatment: a preliminary retrospective study. J Appl Oral Sci. 2005 Mar;13(1):72-7. doi: 10.1590/s1678-77572005000100015. PMID 20944885
- [Background] Dammaschke T, Leidinger J, Schafer E. Long-term evaluation of direct pulp capping--treatment outcomes over an average period of 6.1 years. Clin Oral Investig. 2010 Oct;14(5):559-67. doi: 10.1007/s00784-009-0326-9. Epub 2009 Aug 15. PMID 19685086
- [Background] Matsuo T, Nakanishi T, Shimizu H, Ebisu S. A clinical study of direct pulp capping applied to carious-exposed pulps. J Endod. 1996 Oct;22(10):551-6. doi: 10.1016/S0099-2399(96)80017-3. PMID 9198445
- [Background] Mielke CH Jr, Kaneshiro MM, Maher IA, Weiner JM, Rapaport SI. The standardized normal Ivy bleeding time and its prolongation by aspirin. Blood. 1969;34(2):204-215. Blood. 2016 Aug 25;128(8):1023. doi: 10.1182/blood-2016-06-725127. No abstract available. PMID 27563142
- [Background] Fischer DE. Tissue management: a new solution to an old problem. Gen Dent. 1987 May-Jun;35(3):178-82. No abstract available. PMID 3305151
- [Background] Schroder U. Effect of an extra-pulpal blood clot on healing following experimental pulpotomy and capping with calcium hydroxide. Odontol Revy. 1973;24(3):257-68. No abstract available. PMID 4518199
- [Background] Lemon RR, Steele PJ, Jeansonne BG. Ferric sulfate hemostasis: effect on osseous wound healing. Left in situ for maximum exposure. J Endod. 1993 Apr;19(4):170-3. doi: 10.1016/s0099-2399(06)80681-3. PMID 8326261
- [Background] Nosrat IV, Nosrat CA. Reparative hard tissue formation following calcium hydroxide application after partial pulpotomy in cariously exposed pulps of permanent teeth. Int Endod J. 1998 May;31(3):221-6. doi: 10.1046/j.1365-2591.1998.00147.x. PMID 10321166
- [Background] Mass E, Zilberman U. Clinical and radiographic evaluation of partial pulpotomy in carious exposure of permanent molars. Pediatr Dent. 1993 Jul-Aug;15(4):257-9. No abstract available. PMID 8247900
- [Background] Holland R, de Souza V, de Mello W, Nery MJ, Bernabe PF, Otoboni Filho JA. Permeability of the hard tissue bridge formed after pulpotomy with calcium hydroxide: a histologic study. J Am Dent Assoc. 1979 Sep;99(3):472-5. doi: 10.14219/jada.archive.1979.0317. PMID 112134
- [Background] Witherspoon DE. Vital pulp therapy with new materials: new directions and treatment perspectives--permanent teeth. J Endod. 2008 Jul;34(7 Suppl):S25-8. doi: 10.1016/j.joen.2008.02.030. PMID 18565368
- [Background] Bakland LK, Andreasen JO. Will mineral trioxide aggregate replace calcium hydroxide in treating pulpal and periodontal healing complications subsequent to dental trauma? A review. Dent Traumatol. 2012 Feb;28(1):25-32. doi: 10.1111/j.1600-9657.2011.01049.x. Epub 2011 Sep 5. PMID 21895969
- [Background] Parirokh M, Torabinejad M. Mineral trioxide aggregate: a comprehensive literature review--Part I: chemical, physical, and antibacterial properties. J Endod. 2010 Jan;36(1):16-27. doi: 10.1016/j.joen.2009.09.006. PMID 20003930
- [Background] Barrieshi-Nusair KM, Qudeimat MA. A prospective clinical study of mineral trioxide aggregate for partial pulpotomy in cariously exposed permanent teeth. J Endod. 2006 Aug;32(8):731-5. doi: 10.1016/j.joen.2005.12.008. Epub 2006 Jun 23. PMID 16861071
- [Background] Monteiro Bramante C, Demarchi AC, de Moraes IG, Bernadineli N, Garcia RB, Spangberg LS, Duarte MA. Presence of arsenic in different types of MTA and white and gray Portland cement. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Dec;106(6):909-13. doi: 10.1016/j.tripleo.2008.07.018. Epub 2008 Oct 4. PMID 18835535
- [Background] Santos AD, Moraes JC, Araujo EB, Yukimitu K, Valerio Filho WV. Physico-chemical properties of MTA and a novel experimental cement. Int Endod J. 2005 Jul;38(7):443-7. doi: 10.1111/j.1365-2591.2005.00963.x. PMID 15946264
- [Background] Torabinejad M, Hong CU, McDonald F, Pitt Ford TR. Physical and chemical properties of a new root-end filling material. J Endod. 1995 Jul;21(7):349-53. doi: 10.1016/S0099-2399(06)80967-2. PMID 7499973
- [Background] Belobrov I, Parashos P. Treatment of tooth discoloration after the use of white mineral trioxide aggregate. J Endod. 2011 Jul;37(7):1017-20. doi: 10.1016/j.joen.2011.04.003. Epub 2011 May 28. PMID 21689563
- [Background] Tarbet WJ, Silverman G, Stolman JM, Fratarcangelo PA. Clinical evaluation of a new treatment for dentinal hypersensitivity. J Periodontol. 1980 Sep;51(9):535-40. doi: 10.1902/jop.1980.51.9.535. PMID 6999149
- [Background] Hodosh M, Hodosh SH, Hodosh AJ. Maintenance of pulpal vitality using potassium nitrate-polycarboxylate cement cavity liner. Quintessence Int. 1991 Jun;22(6):495-502. PMID 1882043
- [Background] Hodosh AJ, Hodosh S, Hodosh M. Potassium nitrate-zinc oxide eugenol temporary cement for provisional crowns to diminish postpreparation tooth pain. J Prosthet Dent. 1993 Dec;70(6):493-5. doi: 10.1016/0022-3913(93)90260-u. PMID 8277435
- [Background] Hodosh M, Hodosh SH, Hodosh AJ. Capping carious exposed pulps with potassium nitrate, dimethyl isosorbide, polycarboxylate cement. Dent Today. 2003 Jan;22(1):46-51. No abstract available. PMID 12616888
- [Background] Borissov, S. Tsanova, D. Sivrev. Tissue Response of Dental Pulp in Dogs Following Direct Capping With Potassium Nitrate in Polycarboxylate Cement. Bulgarian Journal of Veterinary Medicine. 2007;10:35-43
- [Background] Tsanova ST, Kundev KK. Dynamics of potassium and nitrate ions release from polycarboxylate cement with 5% KNO3. Folia Med (Plovdiv). 2000;42(2):61-4. PMID 11217288
- [Background] Gudkina J, Mindere A, Locane G, Brinkmane A. Review of the success of pulp exposure treatment of cariously and traumatically exposed pulps in immature permanent incisors and molars. Stomatologija. 2012;14(3):71-80. PMID 23128488
- [Background] Keswani D, Pandey RK, Ansari A, Gupta S. Comparative evaluation of platelet-rich fibrin and mineral trioxide aggregate as pulpotomy agents in permanent teeth with incomplete root development: a randomized controlled trial. J Endod. 2014 May;40(5):599-605. doi: 10.1016/j.joen.2014.01.009. Epub 2014 Mar 6. PMID 24767550
- [Background] Ghoddusi J, Shahrami F, Alizadeh M, Kianoush K, Forghani M. Clinical and radiographic evaluation of vital pulp therapy in open apex teeth with MTA and ZOE. N Y State Dent J. 2012 Apr;78(3):34-8. PMID 22803275
- [Background] El-Meligy OA, Avery DR. Comparison of mineral trioxide aggregate and calcium hydroxide as pulpotomy agents in young permanent teeth (apexogenesis). Pediatr Dent. 2006 Sep-Oct;28(5):399-404. PMID 17036703
- [Background] Kamel M S, Ahmed G M, Yousef H A, AL-Mogy S A. An Improved Technique OF pulp capping by using the Metal Cap with Different Types of Materials. Cairo dental journal .2014;30:1955-1963.